CLINICAL TRIAL: NCT04994756
Title: Stroke Thrombectomy and Aneurysm Registry
Acronym: STAR
Status: Recruiting | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Alejandro Spiotta, Professor-Faculty, Medical University of South Carolina
Other Study IDs: Pro00090704
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Thromboses, Intracranial; Aneurysm, Brain
MeSH Terms: conditions — Stroke; Intracranial Thrombosis; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stroke
  Interventions: Procedure: Stroke/Thrombectomy/Aneurysm-specific surgical procedures
- Thrombectomy
  Interventions: Procedure: Stroke/Thrombectomy/Aneurysm-specific surgical procedures
- Aneurysm
  Interventions: Procedure: Stroke/Thrombectomy/Aneurysm-specific surgical procedures

INTERVENTIONS:
Procedure: Stroke/Thrombectomy/Aneurysm-specific surgical procedures — Participants are retrospectively and/or prospectively entered into registry based on disease indication and respective surgical procedure.

SUMMARY:
This international multi-center registry is used to collect existing information and outcomes for patients undergoing an operation for treatment of injuries to the brain including the blockage of blood flow to an area of the brain, an abnormal ballooning of an artery, abnormal tangling of blood vessels, abnormal formation of blood vessels, tearing of vein, and bleeding in the brain. This information is used to help predict outcomes that undergo an operation for treatment of the above-listed brain injuries. Additionally, the information is used to compare techniques and devices' effects on technical and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgical intervention for central nervous system vascular lesion
* Between 1 and 120 years of age

Exclusion Criteria:

* No exclusion criteria

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patients between 1 and 120 years of age, undergoing surgical intervention for central nervous system vascular lesions.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2055-01-01 (Estimated); Study Completion 2055-01-01 (Estimated)

PRIMARY OUTCOMES:
Post-procedure hemorrhage rate changes | 90 days
  Researchers examine changes in hemorrhage rates in post-stroke patients
Occlusion rates | 90 days
  Measure of how thrombectomy procedure success in relation to reduced occlusion
Complication rates | 90 days
  Measure of post-procedure complication rates in stroke/aneurysm patients
Retreatment rates | 90 days
  Measure of patient retreatment post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Robinson, MS, Study Director — Medical University of South Carolina
Locations (63):
- United States (54):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Loma Linda University, Loma Linda, California
  - Cottage Health Research Institute, Santa Barbara, California
  - Nuvance Health, Danbury, Connecticut
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Health System, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - The Queens Health Center, Honolulu, Hawaii
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Endeavor Health, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Louisiana State University Health Shreveport, Shreveport, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Michigan Health-West, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Rutgers University, New Brunswick, New Jersey
  - Global Neurosciences Institute, Pennington, New Jersey
  - Albany Medical Center, Albany, New York
  - The Feinstein Institutes for Medical Research, Great Neck, New York
  - Stony Brook University, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Raleigh, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Mercy Health, Toledo, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Alleghany Hospital, Pittsburgh, Pennsylvania
  - Geisinger Medical Group, Wilkes-Barre, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - The University of Texas Medical Branch at Galveston, Galveston, Texas
  - Valley Baptist Medical Center, Harlingen, Texas
  - Baylor College of Medicine, Houston, Texas
  - HCA Houston Healthcare Kingwood, Kingwood, Texas
  - Texas Stroke Institute, Plano, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- University of Saskatchewan, Saskatoon, Canada
- Germany (2):
  - Universitätsmedizin Göttingen, Göttingen
  - University Clinic for Neuroradiology, Magdeburg
- Hyogo College of Medicine, Hyōgo, Japan
- Centro Hospitalar Universitário de Lisboa Central, Lisbon, Portugal
- Chonnam National University Hospital, Gwangju, South Korea
- Hospital Universitario La Paz, Madrid, Spain
- Universitätsspital Basel, Basel, Switzerland
- Médica Uruguaya, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No